CLINICAL TRIAL: NCT01620320
Title: Évaluation de l'Echographie de Stress Par Comparaison à la Coronarographie Comme Outil Non Invasif de détection de la resténose Intra endoprothèse du Tronc Commun
Brief Title: Stress Echocardiography Versus Coronary Angiography for Left Main Stenosis Detection
Acronym: ESTRIE-TC
Status: Withdrawn | Type: Observational
Why Stopped: No Funding
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Paul Farand, Doctor, Université de Sherbrooke
Other Study IDs: projet #10-011
Record Dates: First submitted 2010-07-16; First posted 2012-06-15 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Left Main Coronary Artery Disease; Stenosis
Keywords: Left main coronary artery; Coronary artery disease; Stress echography; Intrastent stenosis
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stress echography: Nine to twelve months after their left main angioplasty, patients will go through a stress echo and then the usual control angiography (done routinely in most patient in our center). Patients will act as their own control.
  Interventions: Other: Stress echocardiography

INTERVENTIONS:
Other: Stress echocardiography — Patients able to exercise will have a treadmill test + echography; the others will have a dobutamine echography.
  Other Names: Dobutamine echocardiography; Treadmill echocardiography

SUMMARY:
Left main stenosis use to be treated by bypass but with the improvement of angioplasty techniques, an increasing number of patients are submit to left main coronary angioplasty. Consequences of left main intra stent stenosis can be disastrous yet, for the moment, no precise recommendation concerning the follow up of these patients exist. The investigators ought to determine if stress echocardiography can predict left main intra stent stenosis as well (non inferiorly)as control angiography that use to be done.

DETAILED DESCRIPTION:
All patients of the study will pass coronary angiogram and stress echocardiography (treadmill of dobutamine).

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old able to give consent and having had left main angioplasty.

Exclusion Criteria:

* Bypass on the left anterior descending coronary artery or left circumflex (" protected left main ")
* Treating physician judge that angiography need to be done straightaway
* Follow up elsewhere than the CHUS
* Patient refusal
* Pregnant women
* Stress echo contraindication(Severe high blood pressure or malignant arrhythmia)or condition that limits interpretation (Left bundle branch block or pacemaker rhythm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to teaching hospital or stent from community hospitals to teaching hospital and having left main angioplasty
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between stress echocardiography results for the detection of left main prosthesis stenosis with coronary angiogram results. | 9 to 12 months after left main angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, Cardiologue, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, departement de cardiologie, Sherbrooke, Quebec, Canada